CLINICAL TRIAL: NCT01341678
Title: Circadian Rhythm Modulation by Dietary Phosphorus in Chronic Kidney Disease (CKD)
Brief Title: Circadian Rhythm Modulation by Dietary Phosphorus in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geoffrey Block (Other)
Responsible Party: Sponsor-Investigator, Geoffrey Block, Director of Research, Denver Nephrologists, P.C.
Organization: Denver Nephrologists, P.C. (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: CMD 004
Record Dates: First submitted 2011-04-23; First posted 2011-04-26 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; phosphorus; circadian rhythm; saliva
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Phosphorus Diet (Other): Diet containing 1500mg of phosphorus per day
  Interventions: Other: Diet Only
- Restricted Phosphorus Diet (Other): Diet containing 750mg of phosphorus per day and administration of a phosphate binder (lanthanum carbonate)
  Interventions: Drug: Lanthanum Carbonate
- High Phosphorus Diet (Other): Diet containing 3000mg of phosphorus per day and phosphorus supplementation (NeutraPhos)
  Interventions: Dietary Supplement: NeutraPhos

INTERVENTIONS:
Drug: Lanthanum Carbonate — Diet will be supplemented with 1000mg at each meal
  Other Names: Fosrenol
  Arms: Restricted Phosphorus Diet
Dietary Supplement: NeutraPhos — Diet will be supplemented with NeutraPhos
  Other Names: Phosphorus supplementation
  Arms: High Phosphorus Diet
Other: Diet Only — Diet containing 1500mg of phosphorus
  Arms: Normal Phosphorus Diet

SUMMARY:
The purpose of this study is to describe the circadian rhythm of serum and salivary phosphorus in patients with chronic kidney disease and determine its' modification in response to changes in dietary phosphate load.

DETAILED DESCRIPTION:
In normal healthy individuals, there is a 12-hour and 24-hour circadian rhythm of serum phosphorus (serum P) with a nadir in early-mid morning, a rise to a minor peak in the afternoon (around 4:00PM), and a further rise to a major peak just after midnight. In a study of 6 healthy male patients, Portale et al found that the 12-hour component is modified by dietary P intake whereas the 24-hour rhythm in serum P is independent of the intake of phosphorus. Additionally, this trial demonstrated a large swing in amplitude between peak and nadir serum P in the normal healthy subjects (1.2 mg/dL) and also demonstrated a large difference in mean 24-hour serum P with normal vs. high dietary P intake, however no difference in fasting AM serum P results was observed. These findings may suggest the poor performance of serum P as a biomarker of intervention aimed at P load reductions via treatment options such as phosphate binders or salivary P-binder chewing gum.

While the circadian rhythm of serum phosphorus in healthy individuals has been described, no data exists on the circadian rhythm of salivary P, nor has the circadian rhythm of serum P been described in subjects with moderate kidney disease exposed to various levels of dietary P exposure. In recent years, saliva has been found to be a good indicator of the plasma level of various substances, one of which being phosphorus. Specifically, increased salivary P excretion has been reported in patients with CKD. Daily salivary secretion volume ranges between 500 - 700 mL/day, therefore salivary P has recently been established as a previously unaccounted for source of phosphorus, contributing a conservative estimate of 366 mg/day and 2500 mg/week of immediately bioavailable phosphorus.

There is a significant amount of data available regarding the utilization of serum P as a biomarker of intervention aimed at phosphorus load reductions; however, minimal information regarding the timing of phosphorus measurements (i.e. when serum P is assessed during a 24-hour period) is available. Wolf et al, have demonstrated that despite an 80% reduction in urinary P with dietary P restriction and treatment with P binders over a 2-week period, there was no change in serum P or in FGF-23. However, both biomarkers were sampled once every 3 days over a 2-week period without regard to the time of day. This suggests that single time point measurements of serum P in patients with CKD do not accurately reflect phosphate load. As such, it is plausible that mean 24-hour serum P, or mean 24-hour serum FGF-23 are better markers of phosphorus load in CKD than single measurements.

Additionally, there are no published indicators of 24-hour mean serum P in patients with CKD. It is reasonable that either salivary P or FGF-23 might be optimal predictors. Therefore, this study will examine the 24-hour mean serum P and its relationship to both single and mean salivary P values as well as single and mean FGF-23 values in the controlled setting of specific low, normal and high phosphate diets. This examination and further understanding of mean serum P values and how they relate to the biomarkers of FGF-23 and salivary P with variation in intestinal phosphate load will inform the design and conduct of future interventional trials assessing reductions in phosphorus load.

This study is a single-center, exploratory trial in subjects with reduced kidney function. A total of 9 eligible subjects with an estimated GFR between 30 - 45 mL/min ± 10% and 3 normal healthy subjects as control will be sequentially exposed to three different Phosphorus diets (normal, low and high).

Study assessments will occur in both the inpatient (observation) and outpatient (clinic) setting. A total of four observational inpatient days (Days 7, 12, 18, and 29) will be required throughout the study. Serum, saliva, and urine specimens will be collected at specified time-points beginning at the Day 1 visit and concluding at the Day 36 Follow-Up visit. During the inpatient study visits, blood, urine, and salivary samples will be collected every 4 hours.

Subjects will be provided with specific diets created using a 1500 mg P base diet supplemented with NeutraPhos® to achieve the desired P load as described in the table below. During treatment period 2 (Low P Diet), patients will receive an alternative low P diet and additionally receive lanthanum carbonate 1000 mg with each meal to ensure a low dietary P load.

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years of age
* The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board
* Screening estimated glomerular filtration rate (eGRF) greater than or equal to 30 and less than or equal to 45 mL/min/1.72m2 plus or minus 10% for subjects with CKD and greater than 60mL/min for subjects acting as normal healthy controls
* Willing and able to cooperate with all aspects of the study protocol
* No evidence of significant gastrointestinal (GI) disorder that would impair GI motility or function
* No recent active illness or hospitalization within 12 weeks prior to the Day 1/Baseline visit
* No recent or voluntary change in diet within 4 weeks prior to Day 1/ Baseline visit
* No history of intolerance or adverse effects to lanthanum carbonate
* No use of calcium supplements for at least 2 weeks prior to Day 1
* Must have no dietary restrictions or significant allergies and be willing to eat a non-vegan standardized meal
* Subjects taking nutritional vitamin D or any active vitamin D must be on stable doses with no change during the 4 week period prior to Day 1

Exclusion Criteria:

* Current history of drug or alcohol abuse as assessed by the Principal Investigator
* Receiving active chemotherapy treatment for a malignancy
* Has received dialysis or has acute kidney injury within 12 weeks prior to screening or during screening
* Subject has a clinical condition that in the judgement of the Principal Investigator could potentially pose a health risk to the patient while involved int he study
* Received or has received an investigational product (or is currently using an investigational device) within 30 days prior to screening
* Evidence of active (clinically significant) infections within 14 days prior to Day1/ Baseline visit (in the opinion of the investigator)
* Use of phosphate binding medications (calcium carbonate or acetate with meals, lanthanum carbonate, or sevelamer carbonate)within 7 days prior to the Day 1/ Baseline visit
* Significant GI co-morbidity that would preclude use of lanthanum carbonate phosphate binder (e.g. colostomy with unformed stool, uncontrolled diarrhea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Circadian rhythm of serum phosphorus | 24 hour
  After 1 week of a controlled phosphorus diet patients will be hospitalized for 24 hours and serum phosphorus will be obtained every 4 hours. After a 4 day washout, each subject will cross over to a low phosphorus diet (for 1 week) followed by a 4 day washout and cross over to a high phosphorus diet for 1 week. At the end of each weekly diet a 24 hour hospitalization will occur with samples collected every 4 hours.
Circadian rhythm of plasma fibroblast growth factor 23 (FGF23) | 24 hours
  After 1 week of a controlled phosphorus diet patients will be hospitalized for 24 hours and FGF23 will be obtained every 4 hours. After a 4 day washout, each subject will cross over to a low phosphorus diet (for 1 week) followed by a 4 day washout and cross over to a high phosphorus diet for 1 week. At the end of each weekly diet a 24 hour hospitalization will occur with samples collected every 4 hours.
Circadian rhythm of salivary phosphorus | 24 hours
  After 1 week of a controlled phosphorus diet patients will be hospitalized for 24 hours and salivary phosphorus will be obtained every 4 hours. After a 4 day washout, each subject will cross over to a low phosphorus diet (for 1 week) followed by a 4 day washout and cross over to a high phosphorus diet for 1 week. At the end of each weekly diet a 24 hour hospitalization will occur with samples collected every 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States